CLINICAL TRIAL: NCT03474575
Title: EXADOM: Early Supported Discharge and Enhanced Homecare After Emergency Department Admission for Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Early Supported Discharge and Enhanced Homecare After Emergency Department Admission for Acute Exacerbation of COPD
Acronym: EXADOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38RC16.275
Record Dates: First submitted 2018-02-09; First posted 2018-03-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: COPD
Keywords: homecare, COPD, Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective and Biomedical Research excluding Health Product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD patient (Other): Prevention of re-hospitalization rate for Early supported discharge and enhanced homecare to patient admited for COPD exacerbation
  Interventions: Other: Prevention

INTERVENTIONS:
Other: Prevention — The purpose is to establish a safe and effective way of discharging COPD patients from emergency department by providing enhanced home care.

SUMMARY:
The prevalence of chronic obstructive pulmonary disease (COPD) is between 8 and 15% of the adult population in 2010. This prevalence is expected to increase over the coming decades as the population ages and exposure to the risk factors for the disease continues. The evolution of COPD is marked by the occurrence of exacerbations of varying severity responsible for 1% of emergency department admission. Thus,95% of COPD patients admitted to emergency department for exacerbation are hospitalized.

Several recent studies seem to show that an early discharge from hospital with home care can reduce the rate of rehospitalisation and mortality of COPD patients. These preliminary data on low numbers need to be confirmed. In addition, it seems necessary to identify the phenotypes of patients who benefit most from these early exits.

Exadom project (supported by Rhône-Alpes-Auvergne Regional Health Authorities (ARS), AstraZeneca and Grenoble Alpes University Hospital) aims to establish a safe and effective way of discharging patients by providing enhanced home-based care for AECOPD.

DETAILED DESCRIPTION:
Exadom project (supported by Rhône-Alpes-Auvergne Regional Health Authorities (ARS) , Grenoble Alpes University Hospital) aims to establish a safe and effective way of discharging COPD patients from emergency department by providing enhanced home care.

This program implements ambulatory care immediately after leaving the emergency department with a main goal of reducing hospital readmission during the first month. The home-based support includes daily visits at home conducted by the home care provider's nurses from day 1 to day 7, telephone calls at days 14 and 21 and a final home visit one month after discharge from the emergency department. Blood samples will be collected at inclusion, day 7 and one month during home visit and urine samples at inclusion, day 2, day 4 and one month during home visit .Telephone follow-up at 3, 6 months and one year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Current or former smoker, with at least 10 pack-years
* previous history of COPD with concordant spirometry results
* Admission to the emergency department for an exacerbation defined as an acute event which is characterized by a degradation of respiratory symptoms greater than the usual daily variations and requiring a change in therapeutic management
* Patient with mild exacerbation characterized by a DECAF score at 0 or 1. (DECAF score: Dyspnea, Eosinopenia, Consolidation on chest x-ray, Acidaemia, and atrial Fibrillation. One point for each criterion. Mortality at one month is less than 3% if the DECAF score is 0 or 1).
* Residence within 30km of Grenoble Alps University Hospital
* Patient legally able to give consent
* Person affiliated to a medical insurance

Exclusion Criteria:

* Dementia or non-communicating patient in French language
* Patient unable to call the emergency department at any time in case of sudden worsening
* Pregnancy or breastfeeding woman
* patient under administrative or judicial supervision
* DECAF Score > 1. Patient's with DECAF score > 1 are considered at too high risk of mortality to be managed at home (they are usually hospitalized).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Rate of hospitalizations | 90 days
  number of an hospitalization being an entry in any hospital or clinic , whatever the length of the stay

SECONDARY OUTCOMES:
Rate of all cause of hospitalizations | 6 months and one year
  number of an hospitalization being an entry in any hospital or clinic , whatever the length of the stay for all cause
hospitalization rate for COPD exacerbation aggravation | 3,6 and 12 months
  number of an hospitalization being an entry in any hospital or clinic , whatever the length of the stay for COPD exacerbation aggravation
Hospitalization rate for worsening for cardio-respiratory symptoms | one year
  number of hospitalizations due to myocardial infarction, cardiac failure, stroke
Mortality | 3, 6 and 12 months
  number of death
Determinants of hospitalization | 30 days
  measures of biological and clinical markers collected at baseline and at day 30
Differential of biological and clinical markers | 30 days
  Differential measurements of biological and clinical markers between day 30 and at inclusion
Differential of medical average cost per patient | 3 months
  comparaison between early discharge patient with ambulatory care group and patient with standard care (historical cohort)
Acceptance rate of early ambulatory care | 1 year
  Measured on the basis of a refusal register

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department of University Hospital Grenoble, Grenoble, Auvergne Rhonalpes, France

IPD SHARING:
Plan to Share IPD: No
Not provided